CLINICAL TRIAL: NCT01569386
Title: Low Intensity Physical Activity Leads to Improvement in Brachial-ankle Pulse Wave Velocity in the Affected Leg of Hemiplegics
Brief Title: Low Intensity Physical Activity Leads to Improvement in Brachial-ankle Pulse Wave Velocity of Hemiplegics
Acronym: LIPA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gunma PAZ College (Other)
Collaborators: Kanazawa University (Other)
Responsible Party: Principal Investigator, Akira Kimura,PhD, Professor, Gunma PAZ College
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UMIN000007598
Record Dates: First submitted 2012-03-29; First posted 2012-04-03 (Estimated); Last update posted 2012-04-03 (Estimated); Status verified 2012-04

CONDITIONS: Hemiplegia; Motor Activity; Physical Activity
Keywords: pulse wave velocity; low intensity physical activity; hemiplegia
MeSH Terms: conditions — Hemiplegia; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- low intensity physical activity (Experimental): Daily low intensity physical activity by the half squat
  Interventions: Behavioral: Daily low intensity physical activity by the half squat
- stretch exercise and usual activity (Active Comparator): They do whole body stretch exercise for 20 minute in a day
  Interventions: Behavioral: stretch exercise and usual activity

INTERVENTIONS:
Behavioral: Daily low intensity physical activity by the half squat — They take a meal three times daily. They are a time to do the manual work every day. They watch the TV for two hours every day. And they do a walk of 30 minutes every day. They do a specific exercise. They were trained to conduct 40kcal period(about 20 min.) for adding to the amount of energy consumption of low-intensity physical activity at baseline.Specific exercise that was done the half squat(max knee flexion 70 degree). This squat is carried out in two seconds round trip. This squat is carried out in two seconds round trip. They grab the edge of the table. They put half the weight of the lower limbs paralyzed side. This observer once a week, to record their behavior over 24 hours. Intervention period is up to a maximum of 12 weeks.
  Other Names: low intensity physical activity
  Arms: low intensity physical activity
Behavioral: stretch exercise and usual activity — They take a meal three times daily.They are a time to do the manual work every day.They watch the TV for two hours every day.And they do a walk of 30 minutes every day.They do whole body stretch exercise for 20 minute in a day. An observer once a week, to record their behavior over 24 hours.Their behavior was used to calculate the amount of energy consumption.They are informed of the kcal a day from the viewer.
  Other Names: whole body stretch exercise and usual activity
  Arms: stretch exercise and usual activity

SUMMARY:
Low intensity physical activity by half squat of the elderly people with hemiplegia significantly slow down the pulse wave velocity of the arteries of the lower limbs of the paralyzed side within 8 weeks.

DETAILED DESCRIPTION:
Measurement of aortic pulse wave velocity (PWV) is a noninvasive method for assessing arterial stiffening in atherosclerosis. In hemiplegics, disuse of the affected limb is associated with the muscle wasting leading to development of local atherosclerosis. The brachial-ankle aortic PWV (baPWV) is an indicator of early stage disuse syndrome, and is measured with a device that is particularly useful in elderly hemiplegics.

The LIPA regime was designed to result in an increase of 3.3% (about 40 kcal/day) of daily energy consumption compared to their individual baseline values. This included aerobic exercises and half squats (70° knee flexion) for altogether about 20 minutes, once daily. In addition, the subjects performed passive ankle dorsiflexion-plantar flexion, 30 times/minute for 10 min, once daily. The LIPA was aimed at affecting the passive range of motion in ankle, knee, and hip, and weight bearing on the affected leg in standing position.

ELIGIBILITY:
Inclusion Criteria:

* age above 65 years
* male
* hemiplegic
* onset of stroke within 5 years
* some of them required walking aid indoors
* all of them required a walking aid outdoors

Exclusion Criteria:

* severe functional limitations that precluded any increase in PA
* presence of associated cardiovascular conditions such as uncontrolled hypertension or angina
* presence of undiagnosed or untreated health conditions that manifested as abnormal findings in laboratory test and contraindicated exercise tests

Ages: 65 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 54 (Actual)
Dates: Start 2004-06; Primary Completion 2007-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
brachial- ankle pulse wave velocity(ba-PWV) | Change from Baseline in bar-PWV at 4weeks, 8 weeks and 12weeks
  baPWV were measured using the recently developed device, form ABI/PWV (BP-203RPE; Nihon Colin). This device has four cuffs that can be used to simultaneously measure blood pressure in both arms and both legs, and automatically calculate the ABI. It also records pulse waves with the sensors in the cuffs, computes the difference between transmission time in the arm and transmission time in the ankle, calculates the transmission distance from the right arm to each ankle according to body height, and thus computes the baPWV values from the transmission time and transmission distance.

SECONDARY OUTCOMES:
physical activity levels based on posture and intensity(PIPA), resting heart rate(HR), systolic blood pressure(SBP), ankle-brachial pressure indexABI), heart-aortic pulse wave velocity(ha-PWV) | Change from Baseline in PIPA, ABI, SBP, and HR, ha-PWV, at 4weeks, 8 weeks and 12weeks
  ABI,HR,SBP,ha-PWV were measured using the recently developed device, form ABI/PWV (BP-203RPE; Nihon Colin). This device has four cuffs that can be used to simultaneously measure blood pressure in both arms and both legs, and automatically calculate the ABI. It also records pulse waves with the sensors in the cuffs, computes the difference between transmission time in the arm and transmission time in the ankle, calculates the transmission distance from the right arm to each ankle according to body height, and thus computes the haPWV values from the transmission time and transmission distance.

CONTACTS AND LOCATIONS:
Overall Officials: Akira Kimura, PhD, Study Chair — Gunma PAZ College
Locations (1):
- Gunma PAZ collge, Takasaki, Gunma, Japan

REFERENCES:
- [Background] Kimura A, Miyagi S. A pilot study of advice on physical activity in senior disabled individuals in rural Japan. Asia Pac J Public Health. 2008 Oct;20 Suppl:128-33. PMID 19533871
- See also: Related Info — http://kimuakilabo.main.jp/